CLINICAL TRIAL: NCT05148923
Title: Comparison of Two DCCV Algorithms - Rational Versus Maximum Fixed Energy
Acronym: PROTOCOLENERGY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemocnice AGEL Trinec-Podlesi a.s. (Other)
Responsible Party: Principal Investigator, Lucjan Rucki, Principal Investigator, Nemocnice AGEL Trinec-Podlesi a.s.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IGS202009
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation
Keywords: DCCV; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electric Countershock

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rational energy algorithm (Active Comparator): 150 J, 360 J, 360 J biphasic DCCV
  Interventions: Procedure: Direct current cardioversion (DCCV)
- Maximum fixed energy algorithm (Active Comparator): 3x 360 J biphasic DCCV
  Interventions: Procedure: Direct current cardioversion (DCCV)

INTERVENTIONS:
Procedure: Direct current cardioversion (DCCV) — DCCV is a safe and effective method of treating atrial fibrillation.

SUMMARY:
Direct current cardioversion (DCCV) is a widespread method to restore sinus rhythm in patients with atrial fibrillation. It is a safe and effective method of treating atrial fibrillation. In this study, the investigators want to compare two algorithms. The rational one, with lower initial energy and the second one with the maximum possible shock energy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have atrial fibrillation or atrial tachycardia.
2. Patients must be on therapeutic anticoagulation at least three weeks prior to DCCV or undergo esophageal echocardiography to rule out intracardiac thrombus.
3. Patients come on an empty stomach.
4. Patients must be over 18 years of age.
5. Patients must provide verbal and written informed consent to participate in the study.

Exclusion Criteria:

1. Omitting oral anticoagulant treatment in the last three weeks.
2. Unclear time of onset of palpitations in acute patients without anticoagulation therapy.
3. A different type of arrhythmia than atrial fibrillation or atrial tachycardia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Heart rhythm after DCCV | one minute after DCCV
  sinus rhythm
Incidence of Neurological Adverse Events | two hours after DCCV
  neurological complications

SECONDARY OUTCOMES:
Incidence of skin changes | two hours after DCCV
  none, skin redness, skin burns
Chest pain | one day after DCCV
  0-10 scale of pain severity

CONTACTS AND LOCATIONS:
Overall Officials: Lucjan Rucki, MD, Principal Investigator — Nemocnice AGEL Trinec-Podlesi
Locations (1):
- Nemocnice AGEL Trinec-Podlesi, Třinec, Česká Republika (Česko), Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roman M, Lucjan R, Otakar J, Radim S, Jan C, Radek N, Miroslav H, Libor S, Bogna JG, Jan H, Martin F. Optimizing Energy Delivery in Cardioversion: A Randomized PROTOCOLENERGYTrial of 2 Different Algorithms in Patients With Atrial Fibrillation. Can J Cardiol. 2024 Nov;40(11):2130-2141. doi: 10.1016/j.cjca.2024.06.003. Epub 2024 Jun 8. PMID 38857688